CLINICAL TRIAL: NCT04043611
Title: Effect of Elongation Longitudinaux Avec Decoaption Osteo-Articulaire Exercises in Lumbar Disc Protrusion
Brief Title: Elongation Longitudinaux Avec Decoaption Osteo-Articulaire (ELDOA) in Lumbar Disc Protrusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RiphahIU Nida Rahim Malik
Record Dates: First submitted 2019-08-01; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar Disc Protrusion; ELDOA; Oswestry Disability Index
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative physical therapy management (Active Comparator): Tens and hot pack , Soft tissue mobilization , Maitland's Lumbar segmental mobilization, Traction, Neurodynamics, Active Stretching, McKenzie Prone Extension Exercises
  Interventions: Other: Conservative physical therapy management
- ELDOA (Experimental): Conservative physical therapy management + ELDOA positions
  Interventions: Other: ELDOA

INTERVENTIONS:
Other: Conservative physical therapy management — Tens and hot pack for at least 10 minutes at low back Soft tissue mobilization (Myofascial Release Technique) Maitland's Lumbar segmental mobilization (Grade I & II for pain, Grade III & IV for ROM) Traction (Manual general traction) Neurodynamics (Tensioner technique) Home plan after session (Guided low back exercises):Active Stretching (5-10 repetition with 15-20 second hold), Hamstring, Piriformis McKenzie Prone Extension Exercises
  Arms: Conservative physical therapy management
Other: ELDOA — ELDOA positions (hold for 1 minute,4 alternate days a week) under supervision during session Conservative physical therapy management Tens and hot pack for at least 10 minutes at low back Soft tissue mobilization (Myofascial Release Technique) Maitland's Lumbar segmental mobilization (Grade I & II for pain, Grade III & IV for ROM) Traction (Manual general traction) Neurodynamics (Tensioner technique) Home plan after session (Guided low back exercises):Active Stretching (5-10 repetition with 15-20 second hold),Hamstring,Piriformis
  Arms: ELDOA

SUMMARY:
The aim of this randomized controlled trial will be to determine the effectiveness of ELDOA for treating lumbar disc protrusion. Two randomized groups of patients with lumbar disc protrusion will be treated with conservative physical therapy and the experimental group will be given ELDOA, in addition. Both, male and female patients meeting the inclusion criteria will be included. Patients having concurrent malignancy, infection, trauma or any bony deformity will be excluded

DETAILED DESCRIPTION:
The study is aimed at determining the effects of ELDOA in treating disc protrusion at lumbar region and is being conducted in Max Rehab & Physical Therapy Centre Islamabad and Pakistan Railway General Hospital, Rawalpindi (March 2019-June 2019). Sample size of the study is 34 with confidence interval of 95% and power of 0.8. 30 patients were screened and 29 were included in the study on the basis of inclusion criteria. Sealed envelope contained total 34 questionnaires, 17 for each group. Patients were allocated randomly on the basis of group mentioned on the Performa. Similar conservative rehabilitation protocol was designed for both control and experimental group except for experimental group had ELDOA Exercises in addition. Patients were examined at 1st visit before administration of any treatment and at 4th visit which was also the last one (after completing 4 sessions at alternate days). Baseline evaluation for demographics and symptomatology was taken. Self-reported questionnaire, ODI, NPRS, lumbar ROM and SLR were recorded at first and fourth visit for comparison. 26 patients completed the study while 1 patient from control group and 2 patients from experiment group were lost to follow up and were considered drop outs.

ELIGIBILITY:
Inclusion Criteria:

* Limited ROM (hip/lumbar spine)
* Pain more than 3 on NPRS
* Pain ≥ 3 months

Exclusion Criteria:

* Recurrent disc protrusion
* Spondylolisthesis
* Spondylosis
* Malignancy
* Infection
* Trauma
* Marked bony deformities

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Oswestry disability index | 4th day
  Changes from the Baseline, Oswestry disability index (ODI) was developed in order to assess disability related to pain in individuals with acute, sub-acute, or chronic LBP. The total score of ODI range from 0 (no disability) to 100 (maximum disability). Scores from 0-20 to indicate "minimal disability," 20-40 to indicate "moderate disability," 40-60 to indicate "severe disability," 60-80 to indicate "housebound," and 80-100 to indicate "bedbound". The ODI score is recommended as a back pain-specific measure of disability.
Numeric Pain rating scale | 4th day
  Changes from the Baseline, Numeric Pain rating scale (NPRS) is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain.
Range of Motion (ROM) Lumbar Spine (Flexion) | 4th day
  Changes from the Baseline, ROM of lumbar spine flexion was taken with the help of inclinometer
ROM Lumbar Spine (extension) | 4th day
  ROM of Lumbar spine extension was taken with the help of inclinometer
ROM Lumbar Spine (Right side flexion) | 4th day
  ROM of Lumbar spine right side flexion was taken with the help of inclinometer
ROM Lumbar Spine (left side Flexion) | 4th day
  ROM of Lumbar spine left side flexion was taken with the help of inclinometer
Straight Leg Raising (SLR) | 4th day
  Straight Leg Raising range was taken with the help of inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ghafoor Sajjad, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vroomen PC, de Krom MC, Knottnerus JA. Predicting the outcome of sciatica at short-term follow-up. Br J Gen Pract. 2002 Feb;52(475):119-23. PMID 11887877
- [Background] Peul WC, van den Hout WB, Brand R, Thomeer RT, Koes BW; Leiden-The Hague Spine Intervention Prognostic Study Group. Prolonged conservative care versus early surgery in patients with sciatica caused by lumbar disc herniation: two year results of a randomised controlled trial. BMJ. 2008 Jun 14;336(7657):1355-8. doi: 10.1136/bmj.a143. Epub 2008 May 23. PMID 18502911
- [Background] Tampier C, Drake JD, Callaghan JP, McGill SM. Progressive disc herniation: an investigation of the mechanism using radiologic, histochemical, and microscopic dissection techniques on a porcine model. Spine (Phila Pa 1976). 2007 Dec 1;32(25):2869-74. doi: 10.1097/BRS.0b013e31815b64f5. PMID 18246010
- [Background] Vroomen PC, de Krom MC, Wilmink JT, Kester AD, Knottnerus JA. Diagnostic value of history and physical examination in patients suspected of lumbosacral nerve root compression. J Neurol Neurosurg Psychiatry. 2002 May;72(5):630-4. doi: 10.1136/jnnp.72.5.630. PMID 11971050
- [Background] Fardon DF, Milette PC; Combined Task Forces of the North American Spine Society, American Society of Spine Radiology, and American Society of Neuroradiology. Nomenclature and classification of lumbar disc pathology. Recommendations of the Combined task Forces of the North American Spine Society, American Society of Spine Radiology, and American Society of Neuroradiology. Spine (Phila Pa 1976). 2001 Mar 1;26(5):E93-E113. doi: 10.1097/00007632-200103010-00006. No abstract available. PMID 11242399
- [Background] Kim SH, Kim HS, Kim SW. Lumbar disc herniation in tae kwon do athletic child. J Korean Neurosurg Soc. 2010 Dec;48(6):538-40. doi: 10.3340/jkns.2010.48.6.538. Epub 2010 Dec 31. PMID 21430983
- [Background] Bronfort G, Haas M, Evans R, Leininger B, Triano J. Effectiveness of manual therapies: the UK evidence report. Chiropr Osteopat. 2010 Feb 25;18:3. doi: 10.1186/1746-1340-18-3. PMID 20184717
- [Background] Herzog W. The biomechanics of spinal manipulation. J Bodyw Mov Ther. 2010 Jul;14(3):280-6. doi: 10.1016/j.jbmt.2010.03.004. PMID 20538226
- [Background] Wegner I, Widyahening IS, van Tulder MW, Blomberg SE, de Vet HC, Bronfort G, Bouter LM, van der Heijden GJ. Traction for low-back pain with or without sciatica. Cochrane Database Syst Rev. 2013 Aug 19;2013(8):CD003010. doi: 10.1002/14651858.CD003010.pub5. PMID 23959683
- [Background] Coppieters MW, Andersen LS, Johansen R, Giskegjerde PK, Hoivik M, Vestre S, Nee RJ. Excursion of the Sciatic Nerve During Nerve Mobilization Exercises: An In Vivo Cross-sectional Study Using Dynamic Ultrasound Imaging. J Orthop Sports Phys Ther. 2015 Oct;45(10):731-7. doi: 10.2519/jospt.2015.5743. Epub 2015 Aug 24. PMID 26304637